CLINICAL TRIAL: NCT03766100
Title: The Efficacy of Cognitive Behavioural Therapy for Insomnia (CBT-I) on Sleep in Patients With Rheumatoid Arthritis: the Randomised, Non-blinded, Parallel-group Sleep-RA Trial.
Brief Title: Cognitive Behavioural Therapy for Insomnia on Sleep in Rheumatoid Arthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bente Appel Esbensen (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); Danish Cancer Society (Other); Parker Research Institute (Other)
Responsible Party: Sponsor-Investigator, Bente Appel Esbensen, Researcher Manager, Associate professor, Glostrup University Hospital, Copenhagen
Organization: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-18016081
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis; Insomnia
Keywords: Rheumatoid Arthritis; Insomnia; Sleep; Cognitive Behavioural Therapy for Insomnia; CBT-I; Non-pharmacological treatment; Polysomnography; Actigraphy; Patient reported outcomes
MeSH Terms: conditions — Arthritis, Rheumatoid; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Application of PSG equipment prior to monitoring sleep efficiency and subsequent analysis of results will be conducted by neurophysiology assistants at the Danish Center for Sleep Medicine (DCSM) blinded to participants' allocation. Examination of participants' joints related to the secondary outcome of disease activity will be conducted by a project nurse specialized in rheumatology blinded to participants' allocation. Blood samples related to RA and disease activity will be taken and analysed by a medical laboratory technologist blinded to participants' allocation. Patient Reported Outcome Measures (PROMs) will be collected via questionnaires on tablets handed out by the project manager, who will also conduct the intervention of CBT-I, and therefore not able to be blinded to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Cognitive Behavioural Therapy for Insomnia (CBT-i).
  Interventions: Behavioral: Cognitive behavioural therapy (CBT-i)
- Control group (No Intervention): Insomnia is untreated.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy (CBT-i) — CBT-i aims to alter behaviours that sustain or add to insomnia and correct cognitions that drive these behaviours. The behavioural components of CBT-i are stimulus control (SC) and Sleep Restriction Therapy (SRT). SC works through the extinction of a conditioned arousal that emerges when bed and bedroom have become associated with wakefulness. With SRT time in bed is reduced to build up sleep pressure. When wakefulness is decreased, time in bed is gradually increased until optimal sleep is attained. With the cognitive component, insomnia is treated by identifying and changing unhelpful or inaccurate thinking regarding sleep and distressing emotional responses to insomnia. The last component of CBT-i aims to reduce hyperarousal with relaxation techniques, scheduled worry time, creating a time to unwind, and employing cognitive therapy strategies.
  Arms: Intervention group

SUMMARY:
Introduction:

Rheumatoid arthritis (RA) is a chronic autoimmune inflammatory joint disease that attacks peripheral joints and posterior tissues. More than half of patients with RA also have insomnia, which can modify pain, fatigue, quality of life and comorbidities. Traditional treatment of insomnia is often based on pharmacological drugs, however cognitive behavioural therapy for insomnia (CBT-i) have shown effect in insomnia with less side effects. It remains to determine whether CBT-i can be effective in patients with RA.

The primary objective of this Sleep-RA trial is to assess the efficacy of CBT-i on sleep efficiency in patients with RA at week seven. Key secondary objectives are to estimate the clinical efficacy of CBT-i on wake after sleep onset, total sleep time, sleep onset latency, insomnia, sleep quality, fatigue, RA impact of disease and depressive symptoms at week 26.

Methods & Analysis:

Sleep-RA will be carried out as a randomised controlled trial (RCT) with randomised assignment and two-group parallel design. Patients with RA and insomnia are randomly allocated 1:1 to the intervention group or the control group. The intervention group will once a week for six weeks receive group-based CBT-i, a multi-component intervention of; sleep education, stimulus control, sleep restriction, cognitive therapy and relaxation. The control group will continue treatment as usual (insomnia will remain untreated). Follow-up assessments will be carried out seven and 26 weeks after baseline. The primary outcome is sleep efficiency measured with polysomnography at week seven. Key secondary outcomes are: wake after sleep onset, total sleep time, sleep onset latency, insomnia, sleep quality, fatigue, RA impact of disease and depressive symptoms from baseline to week 26. Polysomnography, actigraphy and Disease Activity Score 28-Joint Count C reactive protein will be assessed by medical staff blinded to group allocation. The project manager will assist the participants with questionnaires and conduct the intervention of CBT-i and will therefore not be blinded to group allocation. With a sample size of 60 patients the trial will have more than 85 % power to detect a mean difference between groups of 6 % points in the primary outcome of sleep efficiency measured at week seven and a reasonable statistical power to explore the clinical efficacy according to the eight key secondary outcome measures at week 26.

Ethics and dissemination:

Ethics approval has been obtained from The Committee on Health Research Ethics. We plan to submit a manuscript with the content of this protocol, and at least one scientific manuscript on the results of the primary and key secondary outcomes to a peer-reviewed journal. Results will be presented at conferences, community and consumer forums and hospital grand rounds.

DETAILED DESCRIPTION:
Introduction:

More than half of patients with rheumatoid arthritis has concomitant insomnia. Insomnia may modify pain, fatigue, quality of life and comorbidities which many patients struggle with. To address this issue, a nurse led sleep outpatient clinic was established in 2015 at the Center for Rheumatology and Spine Diseases in the Capital Region of Denmark. The aim of this clinic is to identify the causes and severity of insomnia in patients with inflammatory joint diseases and to treat it with non-pharmacological initiatives. Eligible patients can be referred to the clinic by rheumatologists and rheumatology nurses. The current project, entitled Sleep-RA, is designed to expand the evidence-based opportunities of non-pharmacological treatment of insomnia within a biopsychosocial perspective among patients with inflammatory joint diseases. First and foremost, we want to assess the efficacy of cognitive behavioural therapy for insomnia on sleep efficiency in patients with rheumatoid arthritis and concomitant insomnia.

Rheumatoid Arthritis:

Rheumatoid arthritis (RA) is a chronic autoimmune inflammatory joint disease (IJD) that affects peripheral joints. The inflammation typically cause tender and swollen joints and cartilage degradation and bone erosions may occur. RA is diagnosed from medical history, physical examination, blood samples and imaging. Prevalence worldwide is 0.4-1.3 % and RA affects women two-three times more frequently than men; onset is most often at 50-60 years of age. The most commonly used method for monitoring disease activity is the Disease Activity Score 28 (DAS28-CRP) based on 28 joint count of tender and swollen joints, C-Reactive Protein (CRP) and 'patient global assessment'. Rheumatological treatment of RA targets reduction of disease activity and is primarily pharmacological with synthetic disease-modifying antirheumatic drugs (csDMARDs), in which methotrexate is the first drug of choice. Biological antirheumatic drugs (bDMARDs) are used in the absence or insufficient effect of csDMARD.

Consequences and symptoms of RA:

Improvements in early diagnosis and medical treatment with antirheumatic drugs, have reduced the incidence of severe joint destruction. However, RA still causes stiffness and swelling in the joints. Some consequences of these symptoms and the inflammation itself are: insomnia, pain, fatigue, reduced physical function, depression and reduced quality of life. About 60-80 % of patients with RA report insomnia compared to 10-30 % in the general population. Patients with RA indicate sleep as one of the most important variables evaluating their medical treatment with antirheumatic drugs, which indicates the impact sleep can have on physical and mental well-being. Pain is also a very common symptom of RA and is associated with fatigue, depressive symptoms, insomnia and inability to work and to cope with social and domestic activities. Furthermore, fatigue is experienced almost universally by individuals with RA while severe fatigue occurs in approximately 50 % of cases. The strongest independent predictors of fatigue are pain, insomnia, depression and physical function. Fatigue is perceived to have a significant impact on physical and social functioning and health care utilization and is a predictor of work dysfunction and overall health status. Pain and fatigue are very important to patient wellbeing and can make the management of other RA symptoms more challenging.

Sleep:

Common definitions of "good" and "bad" sleep in a healthy population are characterised by subjective satisfaction, appropriate timing, adequate duration, high efficiency, and sustained alertness during waking hours. Thus, "sleep health" is seen as a multidimensional pattern of sleep-wakefulness adapted to individual, social, and environmental demands, which promotes physical and mental well-being. These elements are essential to good sleep. To establish a clear meaning of "sleep health", Buysse (2014) has introduced a conceptual model. Five dimensions of sleep were identified as relevant including: sleep duration, sleep continuity or efficiency, timing, alertness/sleepiness, and satisfaction/quality (subjective assessment of good or poor sleep). Within the research field of sleep, studies have mainly focused on negative directions and consequences of sleep and there have been few studies specifically examining the potential benefits of good sleep.

As previously identified, patients with RA suffer from a wide range of disease related consequences and symptoms and most of them can be associated with insomnia. According to observational studies sleep quality is associated with pain, fatigue, quality of life, depression, and disease activity among patients with RA. Insomnia can become long-lasting when the precipitating factor e.g. being diagnosed with a chronic disease as RA to some extend is replaced by perpetuating cognitive and behavioural factors.

Sleep disturbances and cognitive behavioural therapy for insomnia:

The gold standard for identifying insomnia in clinical and research settings is polysomnography (PSG), an objective multi-parametric test. The questionnaires Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI) are the most used and validated questionnaires in assessing patient reported sleep. PSQI has been validated for patients with RA and measures sleep quality and disturbances over the previous month; it differentiates between "good" and "poor" sleepers. Specifically targeting insomnia, the content of ISI corresponds in part to the Diagnostic and Statistical Manual 4th Edition (DSM-IV) diagnostic criteria for insomnia. Actigraphy (small wrist band) is the most valid method to assess sleep/wake behaviour over time (days or weeks).

Insomnia is characterized by difficulty falling asleep or staying asleep as intended and insomnia often leads to inappropriate sleep habits and dysfunctional thoughts related to sleep. Nevertheless, treatment of insomnia is often based on hypnotic drugs that can cause side effects such as tolerance and addiction. In contrast to treatment with hypnotic drugs, cognitive behavioural therapy for insomnia (CBT-i) has demonstrated long-term effects on sleep. So far CBT-i has mostly been tested on people with insomnia and patients with cancer or mental illness with concomitant insomnia. It is a multi-component intervention that aims at teaching patients about health-related significance of sleep and factors that affect it, supporting patients in regulating their sleep habits and dealing with sleep related concerns. CBT-i combines various components: I) stimulus control (e.g. associating the bed and bedroom with sleep), II) sleep restriction (e.g. increasing the homeostatic drive to sleep by reducing time in bed), III) cognitive therapy (i.e. addressing maladaptive beliefs about sleep and reducing arousal and anxiety about sleep and the consequences of not sleeping), IV) sleep hygiene (i.e. establishing behavioural routines to promote restorative sleep) and V) relaxation.

In a recent study in a primary care setting CBT-I conducted as two hours group-based sessions once a week for six weeks with three to eleven participants had significant effect on insomnia. Further, group-based interventions of CBT-i with four to six participants can help break the feeling of isolation.

Rationale:

Even though the prevalence of insomnia is high in patients with RA there have been published results from only very few randomised controlled trials (RCT) in this area. The intervention in most of these studies is based on treatment with hypnotic drugs or other pharmaceutical treatments. Only two studies have been identified as investigating sleep as primary outcome with a non-pharmacological approach, both with physical exercise as intervention. To our knowledge no RCT has yet investigated the effect of CBT-i on insomnia in patients with RA or other (IJD). However, the effect of CBT-i is larger and longer lasting than the effect of pharmaceutical treatments, presumably because patients learn skills they can use to manage sleep at later times. At the Copenhagen Centre for Arthritis Research (COPECARE) the efficacy of high-intensity interval training on sleep in patients with RA has recently been investigated in a pilot/feasibility RCT, data are under review. High-intensity interval training may not appeal to all patients with RA or patients with other IJD. With an intention to offer different non-pharmacological treatments for insomnia in rheumatology outpatient clinics, it is meaningful to assess the efficacy of CBT-i.

CBT-i is often carried out by health professionals with training and experience in psychology. As these professionals rarely are integrated in daily clinical hospital practice, it is difficult to standardize psychologist-led CBT-i in outpatient treatment of insomnia. The clinical effectiveness of group-based CBT-i led by nurses is evidenced in RCTs in European general practice settings.

Previous group-based psychological behavioural interventions, including CBT, have been effective for pain, fatigue, physical function, psychological well-being, social activities and coping resources among patients with RA and CBT-i have had a positive effect on sleep in people with cancer and mental illness.

Aim and objectives:

The aim of Sleep-RA is to assess the efficacy and safety of CBT-i in patients with RA and concomitant insomnia.

Primary objective: To compare the effect of CBT-i relative to a control group on sleep efficiency at week seven in patients with RA and concomitant insomnia.

Key secondary objectives: To compare the effect of CBT-i, relative to a control group, on changes in wake after sleep onset, total sleep time, sleep onset latency, insomnia, sleep quality, fatigue, RA impact of disease and depressive symptoms from baseline to week 26 in patients with RA and concomitant insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA according to American College of Rheumatology/European League Against Rheumatism criteria 2010
* 18 years of age or older
* Patients with low-to-moderate disease activity (DAS28-CRP ≤ 5.1)
* Sleep score ≥ 2 (DANBIO)
* Insomnia severity Index (ISI) ≥ 11
* Unchanged medical treatment with anti-rheumatics > 3 months
* No indication for change of medical treatment with anti-rheumatic drugs the next three months
* Understand and read Danish.

Exclusion Criteria:

* Glucocorticoid administration (i.m., i.a., i.v.) < four weeks
* Oral glucocorticoid administration > 5 mg/day
* Change in oral glucocorticoid dose < three month
* Prior or current contact with rheumatic sleep outpatient clinic
* Night work during the intervention
* Pregnant or breastfeeding
* Current alcohol or drug use disorder
* Patient related circumstances (physical or mental) that impede the ability to give informed consent or adhere to the trial programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Polysomnography (PSG): Sleep efficiency. | Assessed at week 7.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.

SECONDARY OUTCOMES:
Polysomnography (PSG): Wake after sleep onset. | Assessed at week 26.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.
Polysomnography (PSG): Total sleep time. | Assessed at week 26.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.
Polysomnography (PSG): Sleep onset latency. | Assessed at week 26.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.
Insomnia Severity Index (ISI): Insomnia. | Assessed at week 26.
  ISI measures self-reported insomnia severity the last two weeks. ISI is a seven-item questionnaire and each item is rated using a five-point Likert scale ranging from 0 (not at all) to 4 (very much), for a total score ranging from 0 (no insomnia) to 28 (clinical insomnia).
Pittsburgh Sleep Quality Index (PSQI): Sleep quality. | Assessed at week 26.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Bristol Rheumatoid Arthritis Fatigue -Multidimensional Questionnaire (BRAF-MDQ): Fatigue. | Assessed at week 26.
  BRAF-MDQ measures self-reported RA-related fatigue for the previous seven days. It consists of 20 items with four responses ("not at all", "a bit", "part", "much"). Items are combined to create 5 scores, high is worse: Total fatigue score 0-70 Items 1-20 summed, Physical (severity) subscale 0-22 Items 1-4 summed, Living with fatigue subscale 0-21 Items 5-11 summed, Cognitive fatigue subscale 0-15 Items 12-16 summed.
Rheumatoid Arthritis Impact of Disease (RAID): impact of disease. | Assessed at week 26.
  RAID measures self-reported impact of RA on daily life the last seven days. RAID consist of seven items, each item rated using af numerical rating scale (NRS 0-10), high is worse covering pain, physical function, fatigue, sleep, physical well-being, mental well-being and coping. RAID final value = (pain NRS value (range 0-10) x 0.21) + (function NRS value (range 0-10) x 0.16) + (fatigue NRS value (range 0-10) x 0.15) + (physical well-being NRS value (range 0-10) x 0.12) + (sleep NRS value (range 0-10) x 0.12) + (emotional well-being NRS value (range 0-10) x 0.12) + (coping NRS value (range 0-10) x 0.12).
The Hospital Anxiety and Depression Scale for Depression (HADS-D): Depressive symptoms. | Assessed at week 26.
  HADS-D measures self-reported depressive symptoms as psychological morbidity the last seven days. Seven items are rated on a four-point scale and scored from 0-3 with total scores therefore ranging from 0-21. Scores between 0 and 7 represent 'no case', 8 to 10 indicate 'possible case', 11-15 'moderate case' and '15-21' suggest a 'probable severe case of depression'.

OTHER OUTCOMES:
Actigraphy: Sleep efficiency. | Assessed at week 26.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Actigraphy: Wake after sleep onset. | Assessed at week 26.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Actigraphy: Total sleep time. | Assessed at week 26.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Actigraphy: Sleep onset latency. | Assessed at week 26.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Pittsburgh Sleep Quality Index (PSQI): Sleep efficiency. | Assessed at week 26.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Pittsburgh Sleep Quality Index (PSQI): Wake after sleep onset. | Assessed at week 26.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Pittsburgh Sleep Quality Index (PSQI): Total sleep time. | Assessed at week 26.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Pittsburgh Sleep Quality Index (PSQI): Sleep onset latency. | Assessed at week 26.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Disease Activity Score 28-Joint Count C reactive protein' (DAS28-CRP): Disease activity. | Assessed at week 26.
  DAS28-CRP measures disease activity; an objective, reproducible and comparable assessment of the RA activity. A DAS28-CRP greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
28-Joint Count: Tender joints. | Assessed at week 26.
  28-Joint Count measures tender joints by physical examination, reported as yes or no.
28-Joint Count: Swollen joints. | Assessed at week 26.
  28-Joint Count measures swollen joints by physical examination, reported as yes or no.
C-reactive protein level (CRP): Acute-phase reactant value. | Assessed at week 26.
  C-reactive protein level is a blood sample measuring Acute-phase reactant value. Higher value indicate inflammation.
Patients global assessment of disease activity (VAS global patient): patient's global assessment of disease activity. | Assessed at week 26.
  VAS global patient measures patient's self-reported global assessment of disease activity with numerical rating scale (NRS 0-10), high is worse.
Physician's global assessment of the patient's current disease activity (VAS global physician): physician's global assessment of the patient's current disease activity. | Assessed at week 26.
  VAS global physician measures physician's self-reported global assessment of the patient's current disease activity, an overall assessment of how the patient's arthritis is doing with numerical rating scale (NRS 0-10), high is worse.
Bristol Rheumatoid Arthritis Fatigue -Numerical Rating Scale (BRAF-NRS): Fatigue. | Assessed at week 26.
  BRAF-NRS measures self-reported fatigue (severity, coping and effect) the last seven days with numerical rating scale (NRS 0-10), high is worse.
Visual Analogue Scale (VAS pain): Pain. | Assessed at week 26.
  VAS pain measures self-reported current level of RA related pain (VAS 0-100), high is worse.
Multi Dimensional Health Assessment Questionnaire (MDHAQ): Physical function. | Assessed at week 26.
  MD-HAQ measures self-reported physical function the last seven days and contains 10 items covering: dressing, rising, eating, walking, hygiene, reach, grip and everyday activities. Mean of the score = HAQ-score (0,0-3,0), high is worse.
The Short Form [36] Health Survey (SF-36): Health related quality of life. | Assessed at week 26.
  SF-36 measures self-reported health related physical and metal quality of life. SF-36 consists of eight scaled scores, which are the weighted sums of the items in their section. Each scale is transformed into a 0-100 scale. The lower the score the more disability.
Polysomnography (PSG): Sleep efficiency. | Assessed at week 26.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.
Polysomnography (PSG): Wake after sleep onset. | Assessed at week 7.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.
Polysomnography (PSG): Total sleep time. | Assessed at week 7.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.
Polysomnography (PSG): Sleep onset latency. | Assessed at week 7.
  PSG is a multi-parametric test that is used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of the biophysiological changes that occur in the human body when the person is asleep. In Sleep-RA, 17 electrodes are attached to each participant, monitoring: electroencephalogram (EEG), eye movements electro-oculogram (EOG), electromyogram muscle activity or skeletal muscle activation (EMG), heart rhythm (ECG), respiratory airflow, respiratory effort and peripheral pulse oximetry.
Insomnia Severity Index (ISI): Insomnia. | Assessed at week 7.
  ISI measures self-reported insomnia severity the last two weeks. ISI is a seven-item questionnaire and each item is rated using a five-point Likert scale ranging from 0 (not at all) to 4 (very much), for a total score ranging from 0 (no insomnia) to 28 (clinical insomnia).
Pittsburgh Sleep Quality Index (PSQI): Sleep quality. | Assessed at week 7.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Bristol Rheumatoid Arthritis Fatigue -Multidimensional Questionnaire (BRAF-MDQ): Fatigue. | Assessed at week 7.
  BRAF-MDQ measures self-reported RA-related fatigue for the previous seven days. It consists of 20 items with four responses ("not at all", "a bit", "part", "much"). Items are combined to create 5 scores, high is worse: Total fatigue score 0-70 Items 1-20 summed, Physical (severity) subscale 0-22 Items 1-4 summed, Living with fatigue subscale 0-21 Items 5-11 summed, Cognitive fatigue subscale 0-15 Items 12-16 summed.
Rheumatoid Arthritis Impact of Disease (RAID): impact of disease. | Assessed at week 7.
  RAID measures self-reported impact of RA on daily life the last seven days. RAID consist of seven items, each item rated using af numerical rating scale (NRS 0-10), high is worse covering pain, physical function, fatigue, sleep, physical well-being, mental well-being and coping. RAID final value = (pain NRS value (range 0-10) x 0.21) + (function NRS value (range 0-10) x 0.16) + (fatigue NRS value (range 0-10) x 0.15) + (physical well-being NRS value (range 0-10) x 0.12) + (sleep NRS value (range 0-10) x 0.12) + (emotional well-being NRS value (range 0-10) x 0.12) + (coping NRS value (range 0-10) x 0.12).
The Hospital Anxiety and Depression Scale for Depression (HADS-D): Depressive symptoms. | Assessed at week 7.
  HADS-D measures self-reported depressive symptoms as psychological morbidity the last seven days. Seven items are rated on a four-point scale and scored from 0-3 with total scores therefore ranging from 0-21. Scores between 0 and 7 represent 'no case', 8 to 10 indicate 'possible case', 11-15 'moderate case' and '15-21' suggest a 'probable severe case of depression'.
Actigraphy: Sleep efficiency. | Assessed at week 7.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Actigraphy: Wake after sleep onset. | Assessed at week 7.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Actigraphy: Total sleep time. | Assessed at week 7.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Actigraphy: Sleep onset latency. | Assessed at week 7.
  Actigraph is an objective measurement to assess sleep/wake behaviour for several continuous nights. It allows the participant to be mobile and to continue their normal routines while the required data are being recorded in a natural sleep environment. In Sleep-RA actigraph is worn on the non-dominant wrist for one week.
Pittsburgh Sleep Quality Index (PSQI): Sleep efficiency. | Assessed at week 7.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Pittsburgh Sleep Quality Index (PSQI): Wake after sleep onset. | Assessed at week 7.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Pittsburgh Sleep Quality Index (PSQI): Total sleep time. | Assessed at week 7.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Pittsburgh Sleep Quality Index (PSQI): Sleep onset latency. | Assessed at week 7.
  PSQI measures self-reported sleep over the last four weeks. Nine items/18 questions with seven categories, defined with a global sum score for the seven sleep categories differs between good sleep (PSQI global sum score < 5) and bad sleep (PSQI global sum score > 5).
Disease Activity Score 28-Joint Count C reactive protein' (DAS28-CRP): Disease activity. | Assessed at week 7.
  DAS28-CRP measures disease activity; an objective, reproducible and comparable assessment of the RA activity. A DAS28-CRP greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
28-Joint Count: Tender joints. | Assessed at week 7.
  28-Joint Count measures tender joints by physical examination, reported as yes or no.
28-Joint Count: Swollen joints. | Assessed at week 7.
  28-Joint Count measures swollen joints by physical examination, reported as yes or no.
C-reactive protein level (CRP): Acute-phase reactant value. | Assessed at week 7.
  C-reactive protein level is a blood sample measuring Acute-phase reactant value. Higher value indicate inflammation.
Patients global assessment of disease activity (VAS global patient): patient's global assessment of disease activity. | Assessed at week 7.
  VAS global patient measures patient's self-reported global assessment of disease activity with numerical rating scale (NRS 0-10), high is worse.
Physician's global assessment of the patient's current disease activity (VAS global physician): physician's global assessment of the patient's current disease activity. | Assessed at week 7.
  VAS global physician measures physician's self-reported global assessment of the patient's current disease activity, an overall assessment of how the patient's arthritis is doing with numerical rating scale (NRS 0-10), high is worse.
Bristol Rheumatoid Arthritis Fatigue -Numerical Rating Scale (BRAF-NRS): Fatigue. | Assessed at week 7.
  BRAF-NRS measures self-reported fatigue (severity, coping and effect) the last seven days with numerical rating scale (NRS 0-10), high is worse.
Visual Analogue Scale (VAS pain): Pain. | Assessed at week 7.
  VAS pain measures self-reported current level of RA related pain (VAS 0-100), high is worse.
Multi Dimensional Health Assessment Questionnaire (MDHAQ): Physical function. | Assessed at week 7.
  MD-HAQ measures self-reported physical function the last seven days and contains 10 items covering: dressing, rising, eating, walking, hygiene, reach, grip and everyday activities. Mean of the score = HAQ-score (0,0-3,0), high is worse.
The Short Form [36] Health Survey (SF-36): Health related quality of life. | Assessed at week 7.
  SF-36 measures self-reported health related physical and metal quality of life. SF-36 consists of eight scaled scores, which are the weighted sums of the items in their section. Each scale is transformed into a 0-100 scale. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Appel Esbensen, Principal Investigator — Copenhagen Center for Arthritis Research (COPECARE), Center for Rheumatology and Spine Diseases, Rigshospitalet, Denmark.
Locations (1):
- Copenhagen Center for Arthritis Research (COPECARE), Center for Rheumatology and Spine Diseases, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Full dataset to replicate the main analysis will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Abad VC, Sarinas PS, Guilleminault C. Sleep and rheumatologic disorders. Sleep Med Rev. 2008 Jun;12(3):211-28. doi: 10.1016/j.smrv.2007.09.001. PMID 18486034
- [Background] Aletaha D, Smolen JS. Diagnosis and Management of Rheumatoid Arthritis: A Review. JAMA. 2018 Oct 2;320(13):1360-1372. doi: 10.1001/jama.2018.13103. PMID 30285183
- [Background] Edinger JD, Wohlgemuth WK, Radtke RA, Marsh GR, Quillian RE. Cognitive behavioral therapy for treatment of chronic primary insomnia: a randomized controlled trial. JAMA. 2001 Apr 11;285(14):1856-64. doi: 10.1001/jama.285.14.1856. PMID 11308399
- [Background] Davidson JR, Dawson S, Krsmanovic A. Effectiveness of Group Cognitive Behavioral Therapy for Insomnia (CBT-I) in a Primary Care Setting. Behav Sleep Med. 2019 Mar-Apr;17(2):191-201. doi: 10.1080/15402002.2017.1318753. Epub 2017 May 2. PMID 28463015
- [Background] Smith MT, Finan PH, Buenaver LF, Robinson M, Haque U, Quain A, McInrue E, Han D, Leoutsakis J, Haythornthwaite JA. Cognitive-behavioral therapy for insomnia in knee osteoarthritis: a randomized, double-blind, active placebo-controlled clinical trial. Arthritis Rheumatol. 2015 May;67(5):1221-33. doi: 10.1002/art.39048. PMID 25623343
- [Derived] Latocha KM, Loppenthin KB, Ostergaard M, Jennum PJ, Hetland ML, Rogind H, Lundbak T, Midtgaard J, Christensen R, Esbensen BA. The effect of group-based cognitive behavioural therapy for insomnia in patients with rheumatoid arthritis: a randomized controlled trial. Rheumatology (Oxford). 2023 Mar 1;62(3):1097-1107. doi: 10.1093/rheumatology/keac448. PMID 35951745
- [Derived] Latocha KM, Loppenthin KB, Ostergaard M, Jennum PJ, Christensen R, Hetland M, Rogind H, Lundbak T, Midtgaard J, Esbensen BA. Cognitive behavioural therapy for insomnia in patients with rheumatoid arthritis: protocol for the randomised, single-blinded, parallel-group Sleep-RA trial. Trials. 2020 May 29;21(1):440. doi: 10.1186/s13063-020-04282-6. PMID 32471477
- See also: Copenhagen Center for Arthritis Research (COPECARE) — https://www.rigshospitalet.dk/english/departments/centre-of-head-and-orthopaedics/centre-for-rheumatology-and-spine-diseases/copecare/Pages/default.aspx